CLINICAL TRIAL: NCT01675635
Title: A Double-blind, Randomized, Parallel Group Study to Compare the Efficacy and Safety, of Oxycodone Immediate-release Capsules Versus Morphine Immediate-release Tablets in Hospitalized Patients With Moderate to Severe Pain Following Surgery.
Brief Title: OxyNorm Capsules in Post-Operative Pain Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OXYC11-CN-304
Record Dates: First submitted 2012-04-25; First posted 2012-08-30 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OxyNorm Capsules (Experimental): To determine the efficacy and safety of OxyNorm Capsules.
  Interventions: Drug: OxyNorm Capsules
- Morphine tablet (Active Comparator): To determine the efficacy and safety of Morphine tablet.
  Interventions: Other: Morphine tablet

INTERVENTIONS:
Drug: OxyNorm Capsules — dosage:5mg,l0mg and 20mg dosage form:capsule frequency:every 6h, duration:24 hours
  Other Names: OxyNorm
  Arms: OxyNorm Capsules
Other: Morphine tablet — dosage: 10mg and 20mg; dosage form: tablet; frequency: every 6h; duration: 24 hours.
  Other Names: Morphine
  Arms: Morphine tablet

SUMMARY:
The efficacy and safety of oxycodone capsules compared with morphine tablets in hospitalized patients with moderate to severe pain following surgery.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of oxycodone immediate-release capsules compared with morphine immediate-release tablets in hospitalized patients with moderate to severe pain following surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged 18 to 80 years inclusive.
2. Patients who have given written informed consent to participate in the study.
3. Able and willing to communicate with the investigator and his/her staff.
4. Free of anesthesia as assessed through question and answer interaction with nurse at which time oral medication is indicated.
5. Reporting "moderate" or "severe" pain (VAS ≥ 4) related to surgery and requesting analgesics for pain relief.

Exclusion Criteria:

1. Patients have developed tolerance to or dependence on narcotic analgesics and/or alcohol.
2. Patients with ASA ≥ 3 .
3. Have any concomitant medical condition that would be adversely affected by analgesics or confound the quantification of analgesia, or could affect the absorption, metabolism or excretion of the study drugs in any clinically significant fashion.
4. Have known hypersensitivity to any of the study medications or related agents.
5. Have taken analgesic medications within three hours (wash-out) prior to dosing.
6. Have developed complications from the surgical procedure that would confound the study.
7. Have a history of severe iatrogenic adverse experiences.
8. Mothers nursing their infant during the 24 hours following study drug administration, or pregnant women.
9. Patient with Nothing Per Os (NPO) as stated in patient's chart or physician's order.
10. Surgery in patients with epidural anesthesia
11. Patients with Severe impairment of liver at preoperative stage (ALT, AST ≥ 1.5 times upper limit) and abnormal renal function.
12. Patients with medical history of recovering from abnormal surgery anesthesia.
13. Patients with medical history of hypertension (Systolic blood pressure ≥ 180Hg, Diastolic blood pressure 110Hg).
14. Patients with shock.
15. Patients with COPD.
16. According to investigator to determine, patients are in addition the inclusion criteria and exclusion criteria for any other reason than not suitable in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: XinMin Wu, Prof., Principal Investigator — Peking University 1st Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is a randomized, double blind, double dummy, multicenter, parallel group, comparative study to compare the efficacy and safety of oxycodone capsule versus morphine tablet. The subject recruited from hospitalized patients poor with moderate to severe pain following surgery. The duration of the study from 2011 Jul to 2011 Dec.
Pre-assignment Details: There is no run-in or wash out period involved in this study.
  On the protocol 240 subjects was planned to be enrolled, but actually 234 subjects was screened and all randomized. Zero screen failure is reasonable for the indication with this study design.
Groups:
- OxyNorm Capsules: To determine the efficacy and safety of OxyNorm Capsules.
  OxyNorm Capsules: dosage:l0mg dosage form:capsule frequency:every 6h, duration:24 hours
- Morphine Tablet: To determine the efficacy and safety of Morphine tablet.
  Morphine tablet: dosage: 20mg; dosage form: tablet; frequency: every 6h; duration: 24 hours.
Period: Overall Study
Arm/Group | OxyNorm Capsules | Morphine Tablet
Started | 117 | 117
Completed | 117 | 117
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OxyNorm Capsules | Morphine Tablet | Total
Number analyzed (Participants) | 117 | 117 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.44 (11.06) | 43.29 (10.53) | 43.37 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 93 | 194
  Male | 16 | 24 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 116 | 117 | 233
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  China | 117 | 117 | 234
Electrocardiogram test [Count of Participants; unit: Participants] — the judgement of result normal, abnormal non clinical significant or abnormal clinical significant was made by the doctor according to the clinical practice. the study protocol does not have additional or particular requirement.
  Participants
    normal | 88 | 76 | 164
    abnormal, not clinical significant | 29 | 34 | 63
    abnormal,clinical significant | 0 | 5 | 5
America Society of Anesthesiologist classification [Count of Participants; unit: Participants] — ASA Physical Status Classification System
  P1 A normal healthy patient P2 A patient with mild systemic disease P3 A patient with severe systemic disease P4 A patient with severe systemic disease that is a constant threat to life P5 A moribund patient who is not expected to survive without the operation P6 A declared brain-dead patient whose organ are being removed for donor purposes.
  Participants
    P1(Class I) | 61 | 57 | 118
    P2(Class II) | 56 | 60 | 116

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS) in Resting Stage at 6hour (6hour±20 Minutes After Administration of First Dose)
Description: To measure resting VAS at 6h(±20min) after administration of first dose, assessing the intensity of pain, and to conduct inter-group comparison
  Visual Analogue Scale
  0 10 20 30 40 50 60 70 80 90 100
  0 means no pain; 100 means pain as bad as you can image at resting stage
Time Frame: Baseline and 6h (±20min)
Population: 234 subjects in Full Analysis Set (FAS) in which 4 subjects from each group was excluded for Per Protocol(PP) population, so 113 subjects in PP population in each group for the primary endpoint analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- OxyNorm Capsules: To determine the efficacy and safety of OxyNorm Capsules.
  OxyNorm Capsules: dosage: l0mg dosage form:capsule frequency:every 6h, duration:24 hours
Arm/Group | OxyNorm Capsules | Morphine Tablet
Number analyzed (Participants) | 113 | 113
units on a scale
  baseline of Visual Analogue Scale | 46.21 (9.53) | 45.48 (7.94)
  6th hours Visual Analogue Scale | 20.21 (15.66) | 19.94 (15.68)

2. Secondary Outcome: VAS in Both Resting and Coughing Stage at 0.5h, 2h and 24h After Administration of First Dose
Description: To measure the resting and coughing VAS as 0.5h (±5min), 2h (±10min) and 24h (±20min) after administration of first dose, assessing the intensity of pain and to conduct inter-group comparison
Time Frame: Baseline,0.5h (±5min), 2h (±10min) and 24h (±20min)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OxyNorm Capsules | Morphine Tablet
Number analyzed (Participants) | 113 | 113
units on a scale
  Resting baseline of Visual Analogue Scale | 46.21 (9.53) | 45.48 (7.96)
  Resting visual analogue scale before first dose | 46.21 (9.53) | 45.48 (7.96)
  Resting VAS 0.5 hour after first dose | 29.87 (13.59) | 29.80 (12.39)
  Resting VAS 2 hours after first dose | 20.58 (14.40) | 20.89 (12.70)
  Resting VAS 24 hours after first dose | 9.73 (12.52) | 9.75 (11.19)
  Coughing baseline of Visual Analogue Scale | 55.16 (12.15) | 53.91 (10.39)
  Coughing visual analogue scale before first dose | 55.20 (12.12) | 53.91 (10.39)
  Coughing VAS 0.5 hour after first dose | 39.21 (16.56) | 37.96 (13.61)
  Coughing VAS 2hours after first dose | 29.68 (17.91) | 29.30 (13.76)
  Coughing VAS 24hours after first dose | 17.11 (13.51) | 16.27 (12.58)

3. Secondary Outcome: The Use of Rescue Analgesics During the 24-hour Observation Period
Description: To calculate the subject who used rescue analgesics during the 4 dose interval within the 24-hour observation period and to conduct inter-group comparison
Time Frame: 24 hours after the first dose.
Population: in FAS population
Measure: Count of Participants; unit: Participants
Groups:
- Morphine Tablet: To determine the efficacy and safety of Morphine tablet.
  Morphine tablet: dosage:20mg; dosage form: tablet; frequency: every 6h; duration: 24 hours.
Arm/Group | OxyNorm Capsules | Morphine Tablet
Number analyzed (Participants) | 117 | 117
Participants
  First dose interval(0-6h) | 7 | 5
  Second dose interval(7-12h) | 8 | 2
  Third dose interval(13-18) | 1 | 0
  Fourth dose interval(19-24h) | 3 | 2

4. Secondary Outcome: VAS in Coughing Stage at 6h (6h±20min After Administration of First Dose)
Description: To measure coughing VAS at 6h (±20min) after administration of first dose, assessing the intensity of pain, and to conduct inter-group comparison
  Visual Analogue Scale
  0 10 20 30 40 50 60 70 80 90 100
  0 means no pain; 100 means pain as bed as you can image applicable for both resting and coughing stage
Time Frame: Baseline and 6h (±20min)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OxyNorm Capsules | Morphine Tablet
Number analyzed (Participants) | 113 | 113
units on a scale
  Visual Analogue Scale of baseline coughing | 55.16 (12.15) | 53.91 (10.39)
  Visual Analogue Scale after 6hours coughing | 28.81 (17.58) | 28.15 (16.79)

5. Secondary Outcome: Sleeping Quality Assessment
Description: To assess Sleeping quality assessment during 24 hours after administration of first dose and to conduct inter-group comparison
  Sleeping quality scale
  1. Very Good
  2. Good
  3. Fair
  4. Bad
  5. Very Bad
Time Frame: 24 hours after administration of first dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | OxyNorm Capsules | Morphine Tablet
Number analyzed (Participants) | 113 | 113
Participants
  Very Good | 31 | 36
  Good | 38 | 48
  Fair | 38 | 26
  Bad | 5 | 2
  Very Bad | 1 | 1

6. Secondary Outcome: Satisfaction With Pain Control
Description: To assess the Satisfaction with pain control during 24 hours after administration of first dose and to conduct inter-group comparison
  1. Very Satisfied
  2. Satisfied
  3. Fair
  4. Not Satisfied
  5. Not Satisfied at all
Time Frame: 24 hours after administration of first dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Morphine Tablet:: To determine the efficacy and safety of Morphine tablet.
  dosage: 20mg dosage form: tablet; frequency: every 6h; duration: 24 hours.
Arm/Group | OxyNorm Capsules | Morphine Tablet:
Number analyzed (Participants) | 113 | 113
Participants
  Very Satisfied | 38 | 43
  Satisfied | 54 | 58
  Fair | 19 | 12
  Not Satisfied | 2 | 0
  Not Satisfied at all | 0 | 0

7. Secondary Outcome: Comparison of the Total Amount of Study Drugs Used During the 24 Hours
Description: To calculate the total amount of study drugs used during the 24 hours and to conduct inter-group comparison
  The study drug administration is average 6 hours,so the maximal is use 4 times in 24 hours. The investigate to evaluate if the subject need to take the 2nd, 3rd and 4th dose after the mandatory the 1st dose.
Time Frame: 24 hours after administration of first dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | OxyNorm Capsules | Morphine Tablet
Number analyzed (Participants) | 113 | 113
mg | 18.50 (10.37) | 39.82 (21.79)

ADVERSE EVENTS:
Time Frame: The protocol requires safety follow up until 24 hours after the last study medication dosing. So the longest time one subject in the study is 48 hours after the 1st study medication doing, include taking full of the 4 times dosing(intotal 24 hours) following by safety follow up for 24 hours.
Arm/Group | OxyNorm Capsules | Morphine Tablet
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/117
Other Adverse Events (participants affected / at risk) | 35/117 | 35/117
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OxyNorm Capsules (N=117) | Morphine Tablet (N=117)
Nausea (Gastrointestinal disorders) | 15 (15) | 14 (15)
Vomiting (Gastrointestinal disorders) | 7 (7) | 7 (7)
Dizziness (Nervous system disorders) | 7 (7) | 6 (6)
abdominal distension (Gastrointestinal disorders) | 3 (3) | 5 (5)
backache (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
postoperative infection (Infections and infestations) | 2 (2) | 2 (2)
headache (Nervous system disorders) | 2 (2) | 1 (1)
serum creatinine increase (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
alanine aminotransferase increase (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
fever (Infections and infestations) | 1 (1) | 1 (1)
hypertension (Vascular disorders) | 1 (1) | 0 (0)
high tension (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
muculoskeletalache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
expectoration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
epigastric pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
aspartate aminotransferase increase (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
glycosylated hemoglobin derease (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
blood glucose increase (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
leucocyte count increase (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (General disorders) | 0 (0) | 1 (1)
chest uncomfortable (General disorders) | 0 (0) | 1 (1)
blood urea increase (Renal and urinary disorders) | 0 (0) | 2 (2)
swelling (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No